CLINICAL TRIAL: NCT04318925
Title: Evaluation and Follow-up of Patients With Tick-borne Diseases
Brief Title: Evaluation and Follow-up of People With Tick-borne Diseases
Status: Withdrawn | Type: Observational
Why Stopped: No recruitment
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999920030; 20-I-N030
Record Dates: First submitted 2020-03-21; First posted 2020-03-24 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Lyme Disease; Tick-Borne Disease
Keywords: Lyme; Borrelia; Anaplasma; Rickkettsia; Lone Star; Natural History
MeSH Terms: conditions — Lyme Disease; Tick-Borne Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Persons with diagnosed or suspected tick-borne disease age >=18 years

SUMMARY:
Background:

Lyme disease is the most common tick-borne disease in the United States, but other diseases transmitted by ticks have also been on the rise in recent years. Early symptoms of a tickborne disease include fever, headache, fatigue and possible rash. Researchers want to collect information and samples from people with Lyme disease and other tick-borne illnesses to better understand and diagnose these diseases.

Objective:

To evaluate and follow people with tick-borne diseases to help researchers learn more about these infections.

Eligibility:

People ages 18 and older who have or are suspected of having a tick-borne infection.

Design:

Participants will have an initial visit, and visits about 1, 6, and 12 months later. The visits can include a physical exam, blood tests, collection of blood, urine and saliva samples for research, and filling out health-related questionnaires. Participants who have the rash of Lyme disease may be invited to have up to 3 skin punch biopsies of the rash for research.

DETAILED DESCRIPTION:
Lyme disease is a multisystem illness caused by the spirochete Borrelia burgdorferi and it is the most common vector-borne illness in the United States. Tick-borne disease cases reported to the Center for Disease Control and Prevention (CDC) have been on the rise with over 59,000 cases reported in 2017. This protocol is designed to collaborate with University of Maryland School of Medicine for the purpose of recruiting and enrolling patients with Lyme disease and other tickborne illnesses. This is a natural history study which has the objective of developing a rigorously defined population of patients with Lyme disease and other tick-borne illnesses, per CDC case definitions, to serve as the basis for research in multiple aspects of the infections. These research sub-projects have emphasis in exploring the biological markers of tick-borne infections, developing new diagnostic tests for these infections, assessing the clinical course and outcome of patients with these tick-borne infections, and defining the immunological response to the pathogens.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Clinical diagnosis of suspected, confirmed, or probable LB or other TBD per CDC case definitions.
* Has not received antibiotic therapy for tick-borne disease for more than 2 weeks.
* Age >=18 years.
* Able to provide informed consent.
* Subjects must maintain a private physician for non-protocol related medical complaints and for emergency medical treatment required for these or other disorders.

EXCLUSION CRITERIA:

* Post-treatment Lyme disease syndrome
* Women who report they are pregnant.
* Any other condition or history of unacceptably poor compliance that, in the opinion of the investigator, would make the patient unsuitable for enrollment or could interfere with the patient participating in and completing the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary clinical
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Define percentage of participants with suspected, probable, or confirmed TBD, as defined by the CDC case definitions and TBD testing, and measure clinical outcome using established assessment tools and questionnaires. | Assessed annually.
  Identify type of tick-borne disease and clinical outcome.

SECONDARY OUTCOMES:
Utilize current and future technologies to develop new direct and indirect tests and biomarkers for TBDs. These can include, but not limited to, antibody-based testing, antigen-based testing, molecular-based testing, culture. | Ongoing
  Will use samples for developing novel diagnostic testing.
Evaluation of the immune response to the pathogens. These can include, but are not limited to, cytokine testing, cellular response testing, antibody profile, metabolomics, proteomics, transcriptomics, and others. | Ongoing
  Will use samples to explore human immune response to TBDs.
Genomic-based testing for research on pathogen virulence and mutations. | Ongoing
  Will use samples to explore pathogen.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana R Marques, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- University of Maryland Baltimore, Department of Medicine, Baltimore, Maryland, United States

REFERENCES:
- [Background] Nelder MP, Russell CB, Sheehan NJ, Sander B, Moore S, Li Y, Johnson S, Patel SN, Sider D. Human pathogens associated with the blacklegged tick Ixodes scapularis: a systematic review. Parasit Vectors. 2016 May 5;9:265. doi: 10.1186/s13071-016-1529-y. PMID 27151067
- [Background] Coipan EC, Jahfari S, Fonville M, Oei GA, Spanjaard L, Takumi K, Hovius JW, Sprong H. Imbalanced presence of Borrelia burgdorferi s.l. multilocus sequence types in clinical manifestations of Lyme borreliosis. Infect Genet Evol. 2016 Aug;42:66-76. doi: 10.1016/j.meegid.2016.04.019. Epub 2016 Apr 25. PMID 27125686
- [Background] Marques AR. Revisiting the Lyme Disease Serodiagnostic Algorithm: the Momentum Gathers. J Clin Microbiol. 2018 Jul 26;56(8):e00749-18. doi: 10.1128/JCM.00749-18. Print 2018 Aug. PMID 29898997